CLINICAL TRIAL: NCT02290119
Title: PILOT STUDY: Gait and Functional Improvement in Total Knee Arthroplasty With the Use of Verasense for Soft Tissue Balancing: A Randomized, Double-Blind, Controlled Trial
Brief Title: Gait and Functional Improvement in Total Knee Arthroplasty With the Use of Verasense for Soft Tissue Balancing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: as a result of Orthosensor's acquisition by Stryker in July 2018.No final mutually agreed (signed) protocol was found and no clear records of the study data can be retrieved. No accurate and reliable results of this study can be posted.
Sponsor: Orthosensor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 101
Record Dates: First submitted 2014-10-31; First posted 2014-11-13 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis
Keywords: Primary PCL-retaining Total Knee Arthroplasty; Intraoperative Sensors; Ligament Balancing; Clinical Outcomes
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control - Without the use of Verasense (Sham Comparator): Total Knee Replacement without the use of intraoperative sensors
  Interventions: Procedure: Control - Without the use of Verasense
- Sensor-assisted TKR (Verasense) (Active Comparator): Total Knee Replacement with the use of intraoperative sensors
  Interventions: Device: Sensor-assisted TKR (Verasense)

INTERVENTIONS:
Device: Sensor-assisted TKR (Verasense) — Verasense is a single use, disposable device embedded with microelectronics into a standard tibial trial to provide dynamic, intraoperative feedback regarding limb alignment, tibiofemoral position and quantitative pressure at peak contact points in the medial and lateral compartments during total knee replacement surgery. Utilizing sensor-derived data, the surgeon can now evaluate intercompartmental loading throughout the range of motion, and correct for soft-tissue abnormalities while receiving real-time feedback regarding joint balance.
  Arms: Sensor-assisted TKR (Verasense)
Procedure: Control - Without the use of Verasense — Patients in this cohort will undergo manual total knee replacement without the use of Verasense
  Arms: Control - Without the use of Verasense

SUMMARY:
The primary objectives of this study are to understand the effects of soft-tissue balancing on Gait, function and rehabilitation potential after sensor-assisted Total Knee Arthroplasty and correlate Intra-operative subjective feel with OrthoSensor Outputs

Secondary objectives are to quantify and observe:

* Pain medication use
* Swelling
* Muscle strength and girth
* Gait efficiency
* Patient satisfaction
* Activity levels, functional return (i.e., back to work, resume normal activities)
* Patient perception of a balanced knee

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a candidate for a primary PCL retaining total knee arthroplasty
* Subject must be diagnosed with one or more of the following conditions: osteoarthritis, avascular necrosis, rheumatoid or other inflammatory arthritis, post-traumatic arthritis
* Subject is between the age of 45 - 80 years
* Subject is likely to be available for all study visits
* Subject is able and willing to sign the informed consent and follow study procedures

Exclusion Criteria:

* Prior total knee arthroplasty, ligament insufficiencies, prior surgeries such as ACL or PCL reconstructions, posterolateral reconstructions, osteotomies, tibia plateau fractures
* Range of Motion less than 90 degrees, flexion contracture of more than 20 degrees

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Rehabilitation Potential | 6 Months

SECONDARY OUTCOMES:
Knee Society Pain and Functional Scoring (KSS) | 6 month
  The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Forgotten Joint Score (FJS) | 6 month
  The FJS is based on the patients' ability to forget about a joint as a result of the treatment. The FJS assessment is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities.
3D Gait Analysis velocity | 6 Month
  3D gait analysis relates to the range of motion of a joint and the movement velocity. The mean gait speed analysis is considered higher than 1 m/s.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Delanois, MD, Principal Investigator — Sinai Hospital of Baltimore
Locations (1):
- Sinai Hospital of Baltimore - Rubin Institute of Advanced Orthopedics Center for Joint Preservation and Reconstruction, Baltimore, Maryland, United States